CLINICAL TRIAL: NCT06296771
Title: The Effect of a Combined Aerobic and Resistance Exercise (CARE) Training Programme on Cardiometabolic Outcomes in Individuals With Chronic Spinal Cord Injury: A Randomised Controlled Trial
Acronym: CARE training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Chatwalai Sonthikul, PhD student, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345678280233; UBath (Registry Identifier: Chatwalai)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Spinal Cord Injury
Keywords: Chronic spinal cord injury; combined aerobic and resistance exercise training programme; cardiometabolic outcomes; high intensity interval training; resistance training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary energy restriction and exercise group (D+E) (Experimental)
  Interventions: Other: Dietary energy restriction and exercise group (D+E)
- Dietary energy restriction group (D) (Active Comparator)
  Interventions: Other: Dietary energy restriction group (D)

INTERVENTIONS:
Other: Dietary energy restriction group (D) — The participants allocated to the dietary energy restriction group will receive instructions to change their usual dietary intake and maintain their regular physical activity routine for the duration of eight weeks.
  The dietary energy restriction depends on a total calorie deficit of 5000 kcal per week, achieved by the consumption of reduced meal portions. This deficit is computed by subtracting the participants' energy expenditure, as measured by ActiheartTM, rather than relying on reported energy intake. This approach is employed to reduce potential difficulties arising from participants under-reporting their food consumption. The energy deficit is calculated by multiplying the weight of each food item recorded over a 5-day period by an individual factor obtained from energy expenditure data. This calculation enables the determination of the required energy intake for the intervention period.
  Arms: Dietary energy restriction group (D)
Other: Dietary energy restriction and exercise group (D+E) — The individuals within the dietary energy restriction and exercise group will be instructed to reduce their habitual energy intake by 5,000 kcal per week while taking part in physical exercise with a frequency of three sessions per week of HIIT and two sessions per week of resistance exercise throughout a duration of 8 weeks. Sessions can be performed in any order, but we will recommend alternating HIIT and resistance training days and taking the two rest days separately to allow for recovery.
  The exercise programme will start the session by participating in a gentle stretching routine with the objective of reducing the effects of exercise-induced shoulder discomfort. The treatment focuses on the four main muscle groups in the upper body: the latissimus dorsi, the triceps, the rhomboid, the pectoral, and the upper trapezius. Each pose is held in the stretched position for a length of 15 seconds throughout each set, for a total of 4 sets.
  Arms: Dietary energy restriction and exercise group (D+E)

SUMMARY:
The goal of this study is to investigate the effectiveness of an 8-week dietary energy restriction with exercise or dietary energy restriction alone on the cardiometabolic health outcomes of individuals with chronic spinal cord injury. This study is a randomised controlled trial conducted at a single centre, consisting of two parallel arms. The main questions it aims to answer are:

1. the effectiveness of an 8-week dietary energy restriction with exercise or dietary energy restriction alone on cardiometabolic disease biomarker outcomes in individuals with chronic SCI
2. the effectiveness of an 8-week dietary energy restriction with exercise or dietary energy restriction alone on fitness and health outcomes.

Twenty-one participants will be randomly assigned in a 2:1 allocation ratio. The participants will be assigned to either the dietary energy restriction and exercise group (D+E) group, which combines dietary energy restriction and exercise intervention, or the dietary energy restriction group (D) group, which just undergoes dietary energy restriction using sealed envelopes.

DETAILED DESCRIPTION:
This study is a randomised controlled trial conducted at a single centre, consisting of two parallel arms. The recruitment of 21 people with a chronic spinal cord injury will begin through the distribution of advertisements across several channels, including national disability charity websites, internet forums, and social media networking sites. Interested potential participants will be asked to contact the principal researcher for further information via email or telephone correspondence. The principal researcher will email a participant information sheet and health screening questionnaire and conduct a follow-up phone call >48 hours after the participant expresses their initial interest to fully explain what the trial entails and answer any questions. If the potential participant indicates that they wish to take part in the study, the first visit will be scheduled. On the first visit, participants will be asked to provide written informed consent. The study will involve a total of 2 assessment visits (~5 hours each), which will take place before and after an 8-week intervention. For these visits, participants will be asked to arrive after an overnight fast (>10 hours). During these visits, we will first assess anthropometrics by dual-energy X-ray absorptiometry and peripheral quantitative computed tomography. A principal researcher will adipose tissue biopsy by procedure known as 'needle aspiration' and insert a cannula into a vein in the forearm to allow regular blood samples to be taken for 2 hours following the oral consumption of glucose drinks. During the 2-hour glucose test, participants will be asked to complete two questionnaires on pain, and quality of life. Participants will then be given lunch and asked to perform a maximal exercise test on an arm-crank ergometer, muscular strength by hand-held dynamometer, and balance by functional reach test. Participants will be asked to wear a physical activity monitor for 5 days following the initial visit and in the final week of the 8-week period. Participants will also be asked to complete a questionnaire about the satisfaction and perceived benefits of the programme intervention on week 8. After baseline testing, eligible consenting participants will be randomly allocated (2:1) to a dietary energy restriction with exercised (D+E) or dietary energy restriction alone (D) using a sealed envelope and balance groups for key characteristics (age, sex, and and level of injury) at baseline. The participants allocated to the D group will receive instructions to reduce meal portions for a total calorie deficit of 5000 kcal per week and maintain their regular physical activity routine for the duration of eight weeks. This deficit is computed by subtracting the participants' energy expenditure, as measured by ActiheartTM. The individuals within the D+E group will be instructed to reduce their habitual energy intake by 5,000 kcal per week while taking part in physical exercise with a frequency of three sessions per week of HIIT and two sessions per week of resistance exercise throughout a duration of 8 weeks. Throughout the exercise training sessions, participants will receive instructions to employ a chest-worn heart rate (HR) monitor.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for participation in this study are that patients have a chronic SCI that occurred at least one year before, an age range between 18 and 65 years, and sufficient upper limb function to engage in the exercise intervention. Participants must self-report that they use a wheelchair for the majority of their waking hours, namely 75% of their day, and have continually maintained a stable weight within a range of ± 3 kg over the duration of the previous three months.

Exclusion Criteria:

The study will exclude participants who have provided information about their medical conditions, such as unresolved pressure sores, urinary tract infections, active medical conditions that may be a contraindication to exercise testing (ACSM Exercise Testing Guidelines), or current musculoskeletal symptoms of the upper extremities. Individuals who have self-reported the use of medication for type 2 diabetes or pharmaceuticals that influence glucose metabolism will be excluded from involvement in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-05-22 (Estimated); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 8 weeks
  Blood sample
Fasting insulin concentration | 8 weeks
  Serum insulin concentration
Insulin sensitivity | 8 weeks
  Serum insulin concentration

SECONDARY OUTCOMES:
Resting matabolic rate | 8 weeks
  Measured using indirect calorimetry
Body mass | 8 weeks
  Measured using electronic wheelchair scales
Waist and hip circumference | 8 weeks
  Measured using a non-metallic tape
Height | 8 weeks
  Measured using a non-metallic tape
Total body fat percentage | 8 weeks
  Measured using duel-energy x-ray absorptiometry
Total Fat-Free Mass | 8 weeks
  Measured using duel-energy x-ray absorptiometry
Visceral Adipose Tissue | 8 weeks
  Measured using duel-energy x-ray absorptiometry
Total Fat Mass | 8 weeks
  Measured using duel-energy x-ray absorptiometry
Muscle, adipose and bone cross-sectional areas around the tibia and femur | 8 weeks
  Measured using Peripheral quantitative computed tomography
Bone geometry and tissue densities around the tibia and femur | 8 weeks
  Measured using peripheral quantitative computed tomography
adipose tissue | 8 weeks
  Measured using adipose tissue biopsy
Upper extremity muscle strength | 8 weeks
  Handheld dynamometer
Balance | 8 weeks
  The Modified Functional Reach Test
Health-related quality of life | 8 weeks
  Measured using a validated questionnaire
Shoulder Pain | 8 weeks
  Measured using a validated questionnaire
Energy intake and dietary macronutrient composition | 8 weeks
  Estimated using a 5-day weighed food diary
Energy expended in different physical activity intensities (MET categories) (kJ or kcal) | 8 weeks
  Energy expended in different physical activity intensities across 5-days (MET categories) (kJ or kcal)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided